CLINICAL TRIAL: NCT03910699
Title: Uni-center, Patient-blinded, Randomized, 12 Month, Parallel-group, Non-inferiority Study to Compare Outcomes of Three-row Versus Two-row Circular Staplers for Colorectal Anastomosis Formation After Low Anterior Resection for Rectal Cancer
Brief Title: THREE-row Circular STAPLER in Low Anterior Resection for Rectal Cancer
Acronym: THREESTAPLER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Collaborators: Meril Life Sciences Pvt. Ltd. (Industry); I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Inna Tulina, Head of Oncologic Colorectal Surgery Department, Clinic of Colorectal and Minimally Invasive Surgery, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSCS-Z0836
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Anastomotic Leak; Anastomotic Haemorrhage; Anastomotic Complication; Rectal Neoplasms; Staple Misfire; Anastomosis; Anastomotic Stenosis
Keywords: Anastomosis; Anastomotic leakage; Rectal cancer; Total mesorectal excision; Low anterior resection; Anastomotic leak; Colorectal anastomosis; Three-row stapler
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two-row anastomosis (Active Comparator): Colorectal anastomosis is created with a two-row circular surgical stapler
  Interventions: Device: Two-row circular stapler
- Three-row anastomosis (Experimental): Colorectal anastomosis is created with a three-row circular surgical stapler
  Interventions: Device: Three-row circular stapler

INTERVENTIONS:
Device: Three-row circular stapler — Para-aortic lymph node dissection, inferior mesenteric artery skeletonisation and ligation below left colic artery origin, nerve-preserving total mesorectal excision, rectum division with a linear stapler, sigmoid colon division and circular stapler envil fixation with a purse-string suture, end-to-end colorectal anastomosis creation with a three-row circular stapler, defunctioning colostomy is performed.
  Other Names: MirusTM Disposable Circular Stapler 3 Row 29 (MCS-29R3)
  Arms: Three-row anastomosis
Device: Two-row circular stapler — Para-aortic lymph node dissection, inferior mesenteric artery skeletonisation and ligation below left colic artery origin, nerve-preserving total mesorectal excision, rectum division with a linear stapler, sigmoid colon division and circular stapler envil fixation with a purse-string suture, end-to-end colorectal anastomosis creation with a two-row circular stapler, defunctioning colostomy is performed.
  Other Names: Ethicon 29mm Curved Intraluminal Stapler (CDH29A)
  Arms: Two-row anastomosis

SUMMARY:
This trial aims to assess safety and efficacy of three-row circular staplers compared to two-row surgical stapllers in short-term and long-term perspective in patients with rectal cancer undergoing low anterior resection with stapled colorectal anastomosis. All the patients will undergo a low anterior resection. In a half of patients a colorectal anastomosis will be created with a three-row surgical circular stapler. In another half of patients a colorectal anastomosis will be created with a two-row surgical circular stapler.

DETAILED DESCRIPTION:
A low anterior resection for rectal cancer in most cases results in creating a colorectal anastomosis with a surgical circular stapler device. Using a disposable circular stapler with two rows of staples is standard of care nowadays. Colorectal anastomosis dehiscence and subsequent anastomotic leak in postoperative period happens in 5-25% of cases and is a major and life-threatening complication. Thus different improvements to the procedure of creating a colorectal anastomosis are being proposed. One of them is utilizing a three-row instead of a two-row surgical circular stapler.

A three-row surgical stapler has recently been registered and approved for clinical use in Russia. The primary purpose of this study is to find out the rate of colorectal anastomosis leakage when using a three-row circular stapler and to demonstrate that it is at least not bigger than the rate of colorectal anastomosis leakage when using a two-row circular stapler.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated consent to comply with all study procedures and availability for the duration of the study
3. Male or female
4. For females of reproductive potential: not pregnant at the time of screening
5. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
6. Histologically proven primary rectal adenocarcinoma located within 5 to 15 cm from anal verge not involving internal and/or external sphincter muscle

Non-inclusion Criteria:

1. Current use of antiplatelet drugs, acetylsalicylic acid or anticoagulants within 7 days prior to intervention
2. Unresectable tumour, inability to perform a TME with colorectal anastomosis, inability to complete R0 resection or presence of T4b tumour necessitating a multi-organ resection
3. Inability to save the left colic artery
4. Diameter of rectal lumen is unable to contain the working part of the stapler
5. Infection requiring antibiotic treatment within 30 days prior to intervention
6. Anal incontinence prior to surgery (Wexner Continence Grading Scale >=10)
7. Significant comorbidities - ASA > III

Exclusion criteria:

1. Patient lost for observation
2. Inability to complete all the trial procedures
3. Death due to causes unrelated to anastomotic leak in early postoperative period

8. Current smoker or tobacco use within <specify timeframe> 9. Patient wants to withdraw from the clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate | 6 weeks
  The rate of colorectal anastomosis dehiscence documented with an X-ray and/or CT scan

SECONDARY OUTCOMES:
Operating time | 1 day
  The duration of surgical procedure in minutes
Circular stapler misfunction rate | 1 day
  The rate of circular stapler inability to create a colorectal anastomosis in a way declared by the manufacturer
Anastomotic bleeding rate | 30 days
  The rate of bleeding from the line of stapled anastomosis verified by proctoscopy
Re-intervention rate | 6 weeks
  The rate of repeat surgeries due to anastomotic leakage
Early postoperative complications rate | 30 days
  The rate of complications in first 30 days after surgery
The postoperative hospital stay | 1 month
  The number of days from the first day after operation to discharge
Complications of defunctioning stoma | 3 months
  The rate of complications related to defunctioning stoma
Overall quality of life | 7 days before surgery, 1 month, 3 months, 6 months and 12 months after surgery
  Assessed with patient-reported questionnaire SF-36. A total score in each of 8 sections will be calculated and transformed into a 0-100 scale with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disability
Cancer-related quality of life | 7 days before surgery, 1 month, 3 months, 6 months and 12 months after surgery
  Assessed with patient-reported questionnaire EORTC QLQ-C30 with supplementary module EORTC QLQ-CR29. A total score in each of 4 modules (functional scale, global health status, symptom scale, colorectal cancer module) will be calculated and transformed into a 0-100 scale. For Functional scale, Global health status scale and Colorectal cancer module a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. For Symptom scale a score of 100 is equivalent to maximum disability and a score of 0 is equivalent to no disability.
Manifestation of Low Anterior Resection Syndrome (LARS) | 7 days before surgery, 1 month, 3 months, 6 months and 12 months after surgery
  Assessed with patient-reported questionnaire LARS, total score will be calculated (min 0, max 42) for each patient and also each patient will be assigned to either "no LARS" group (total score 0-20), or "minor LARS" group (total score 21-29) or "major LARS" group (total score 30-42)
Adverse events rate | 12 months
  The rate of adverse events related to circular stapler usage
Serious adverse events rate | 12 months
  The rate of serious adverse events related to circular stapler usage

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, MD, Study Director — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally Invasive Surgery - I.M. Sechenov First Moscow State Medical University, Moscow, Russia

REFERENCES:
- [Derived] Nekliudov NA, Tsarkov PV, Tulina IA. Uni-center, patient-blinded, randomized, 12-month, parallel group, noninferiority study to compare outcomes of 3-row vs 2-row circular staplers for colorectal anastomosis formation after low anterior resection for rectal cancer. Medicine (Baltimore). 2019 Jun;98(24):e15978. doi: 10.1097/MD.0000000000015978. PMID 31192938